CLINICAL TRIAL: NCT01613053
Title: Continuation of Drug Supply in Chinese Patients After CAMN107DBR01study Termination
Acronym: MACS2226
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107DCN03
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Gastrointestinal Stromal Tumor
Keywords: Gastrointestinal Stromal Tumor, GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Glivec — 800 mg per day

SUMMARY:
Continuation of drug supply in Chinese patients after CAMN107DBR01study termination.

DETAILED DESCRIPTION:
Five patients who are on treatment of imatinib and deriving clinical benefit after CAMN107DBR01 study termination and written informed consent obtained will enter the trial, all five patients will receive Glivec (8oomg per day) treatment until tumor progression [by RECIST guidelines, version 1.0], unacceptable toxicity, death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Five patients who are on treatment of imatinib and deriving clinical benefit after CAMN107DBR01 study termination and written informed consent obtained.

Exclusion Criteria:

* N/A.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhong, M.D., Principal Investigator — Ruijin Hospital of Shanghai Jiaotong University
Locations (3):
- China (3):
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Guangzhou
  - Novartis Investigative Site, Shanghai